CLINICAL TRIAL: NCT00643149
Title: A Multicenter, Randomized, Double-Blind, Double-Dummy Comparative Trial Of Azithromycin SR Versus Amoxicillin For The Treatment Of Group A Β-Hemolytic Streptococcal Pharyngitis/Tonsillitis In Children
Brief Title: A Multicenter, Randomized, Double-Blind, Double-Dummy Study Of Azithromycin SR Versus Amoxicillin For The Treatment Of Strep Throat In Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A0661071
Record Dates: First submitted 2008-03-19; First posted 2008-03-26 (Estimated); Last update posted 2011-05-17 (Estimated); Status verified 2011-05

CONDITIONS: Tonsillitis
MeSH Terms: conditions — Tonsillitis | interventions — Amoxicillin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: amoxicillin
- 2 (Experimental)
  Interventions: Drug: azithromycin SR

INTERVENTIONS:
Drug: amoxicillin — 10 day regimen, 45 mg/kg/day, given in divided doses every 12 hours
  Arms: 1
Drug: azithromycin SR — 60 mg/kg dose of azithromycin SR was as safe and effective as a 10-day regimen of amoxicillin when used to treat children with strep throat
  Arms: 2

SUMMARY:
The objective was to determine if a single 60 mg/kg dose of azithromycin SR was as safe and effective as a 10-day regimen of amoxicillin (45 mg/kg/day, given in divided doses every 12 hours) when used to treat children with strep throat.

ELIGIBILITY:
Inclusion Criteria:

Patients who had evidence of acute pharyngitis/tonsillitis based on erythematous pharyngeal mucosa or thick exudate covering the pharynx and tonsillar area, and at least one of the following signs or symptoms were included: sore/scratchy throat; pain on swallowing; chills and/or fever cervical adenopathy; scarlet fever rash on the face and skin folds, or red tongue with prominent papillae ("strawberry tongue"). Subjects were required to have a positive rapid antigen detection test (RADT) or a positive culture of the pharynx or tonsils for GABHS.

Exclusion Criteria:

Patients were excluded if they had previously diagnosed disease(s) of immune function or treatment with any systemic antibiotic within the previous 7 days.

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 693 (Actual)
Dates: Start 2003-05; Study Completion 2004-03 (Actual)

PRIMARY OUTCOMES:
Bacteriologic response (eradication or persistence) at the Test of Cure (TOC) visit in the Bacteriologic Per Protocol population | TOC visit (Day 24-28)

SECONDARY OUTCOMES:
Bacteriologic eradication rate at the Long-Term Follow-Up (LTFU) visit | LTFU Visit (Day 38-45)
Clinical response (clinical cure or failure) at the TOC visit in the Bacteriologic Per Protocol population | TOC Visit (Day 24-28)
Clinical response (cure or relapse) at the LTFU visit | LTFU Visit (Day 38-45)
Pathogen susceptibility versus bacteriologic response | Not reported
Adverse events (AEs) were assessed for all treated subjects | Continuous
Vital signs and physical examinations were recorded | Baseline and as necessary
Clinical laboratory testing (hematology and blood chemistry) | As necessary
Azithromycin serum concentrations were determined for patients who vomited within 30 minutes of receiving their azithromycin SR/placebo dose | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (36):
- United States (23):
  - Pfizer Investigational Site, Hoover, Alabama
  - Pfizer Investigational Site, Pelham, Alabama
  - Pfizer Investigational Site, Fresno, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, Evansville, Indiana
  - Pfizer Investigational Site, Newburgh, Indiana
  - Pfizer Investigational Site, Wichita, Kansas
  - Pfizer Investigational Site, Bardstown, Kentucky
  - Pfizer Investigational Site, Springfield, Kentucky
  - Pfizer Investigational Site, Kalamazoo, Michigan
  - Pfizer Investigational Site, Endwell, New York
  - Pfizer Investigational Site, Raleigh, North Carolina
  - Pfizer Investigational Site, Beachwood, Ohio
  - Pfizer Investigational Site, Chesterland, Ohio
  - Pfizer Investigational Site, Cleveland, Ohio
  - Pfizer Investigational Site, Willoughby, Ohio
  - Pfizer Investigational Site, Youngstown, Ohio
  - Pfizer Investigational Site, McMurray, Pennsylvania
  - Pfizer Investigational Site, Pittsburgh, Pennsylvania
  - Pfizer Investigational Site, Bryan, Texas
  - Pfizer Investigational Site, Lake Jackson, Texas
  - Pfizer Investigational Site, Salt Lake City, Utah
  - Pfizer Investigational Site, West Jordan, Utah
- Canada (4):
  - Pfizer Investigational Site, Calgary, Alberta
  - Pfizer Investigational Site, Coquitlam, British Columbia
  - Pfizer Investigational Site, Winnipeg, Manitoba
  - Pfizer Investigational Site, Saskatoon, Saskatchewan
- Costa Rica (4):
  - Pfizer Investigational Site, Escazú, Provincia de San José
  - Pfizer Investigational Site, San José, Provincia de San José
  - Pfizer Investigational Site, Uruca, Provincia de San José
  - Pfizer Investigational Site, San José
- Pfizer Investigational Site, Guatemala City, Departamento de Guatemala, Guatemala
- India (4):
  - Pfizer Investigational Site, Hyderabad, Andhara Pradesh
  - Pfizer Investigational Site, Bangalore, Karnataka
  - Pfizer Investigational Site, Kochi, Kerala
  - Pfizer Investigational Site, Mumbai, Maharashtra

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0661071&StudyName=A%20Multicenter%2C%20Randomized%2C%20Double-Blind%2C%20Double-Dummy%20Study%20Of%20Azithromycin%20SR%20Versus%20Amoxicillin%20For%20The%20Treatment%20Of%20Strep%20Throat%20In